CLINICAL TRIAL: NCT00745381
Title: Gastroenteropancreatic and Unknown Primary Neuroendocrine Registry A Collection of Clinical and Epidemiologic Data Combined With Tissue and Blood From Patients With a Diagnosis of Neuroendocrine Tumors
Brief Title: A Collection of Clinical and Epidemiologic Data Combined With Tissue and Blood From Patients With a Diagnosis of Neuroendocrine Tumors
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 08-105
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Gastric Cancer; Pancreatic Cancer
Keywords: PANCREAS; STOMACH; Questionnaire; 08-105
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All participants will be invited to provide a DNA (blood sample) and tissue sample for the purposes of developing a tissue repository. Blood samples will be collected. Expected accrual is 150 patients per year. Patients who donate blood and/or tissue samples are considered evaluable for protocol; however, it is preferred that both are obtained.

GROUPS / COHORTS (1):
- 1: This registry will be open to all patients with GEPNET or NET of unknown primary.
  Interventions: Other: questionnaire, Blood specimens

INTERVENTIONS:
Other: questionnaire, Blood specimens — All participants will complete an epidemiology study questionnaire as well as a quality of life questionnaire. They will also be asked to donate blood samples. We will request participation in a tissue repository consisting of fresh frozen or paraffin embedded tissue. The repository will be of serum, plasma and tumor tissue. Follow-up will occur on patients every 6 months for the first year after consent and then annually.

SUMMARY:
The purpose of this study is to establish a neuroendocrine tumor registry. A registry is a collection of information. To create this registry, the investigators would like to get information, blood and tumor samples from people with neuroendocrine tumors. By collecting this information and material, the investigators are hoping to learn more about the genetic causes of neuroendocrine tumors. All of this will help us to better understand neuroendocrine cancer, so the investigators can find better ways to treat and diagnose this disease. DNA will be taken from the blood samples and will be used in future studies. This will be an important resource from which the investigators can study genes that may be related to a higher risk of neuroendocrine tumors.

The information collected will include medical information, family history of cancer and your answers to questions about how the cancer affects quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gastroenteropancreatic neuroendocrine tumors or neuroendocrine tumors of unknown primary
* Willing to donate blood samples
* >= 18years old
* Patients may have received prior hormonal therapy, cytotoxic therapy, irradiation, immunotherapy or surgical therapy

Exclusion Criteria:

* Have any condition, which in the opinion of the primary MSKCC clinician or investigators precludes their ability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with GEPNET or NET of unknown primary
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2008-08; Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
To develop a tissue, serum, plasma and DNA bank from individuals with NET. This bank will be combined with epidemiologic and clinical information to create a NET database. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Diane Reidy-Lagunes, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan-Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm